CLINICAL TRIAL: NCT04171531
Title: Treatment for Mixed Urinary Incontinence: Mid-urethral Sling vs. Botox A
Brief Title: Sling vs Botox for Mixed Incontinence
Acronym: MUSA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NICHD Pelvic Floor Disorders Network (Network)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Women and Infants Hospital of Rhode Island (Other); Duke University (Other); University of Pennsylvania (Other); University of Pittsburgh (Other); University of California, San Diego (Other); Kaiser Permanente (Other); University of Texas Southwestern Medical Center (Other); University of Alabama at Birmingham (Other); RTI International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PFDN-31P01; U24HD069031-06 (NIH); UG1HD069013-06 (NIH); UG1HD041267-18 (NIH); UG1HD069010-07 (NIH); UG1HD069006-07 (NIH); UG1HD041261-17 (NIH); UG1HD054214-12 (NIH); UG1HD054241-12 (NIH)
Record Dates: First submitted 2019-11-18; First posted 2019-11-21 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Urinary Incontinence, Stress; Urinary Incontinence, Urge
Keywords: urinary incontinence; midurethral sling; Botulinum toxin A (Botox A ®)
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence, Urge; Urinary Incontinence | interventions — Botulinum Toxins, Type A; Suburethral Slings

STUDY DESIGN:
Intervention Model Description: At 6 months, the effect of treatment with Botox A or mid-urethral sling will be evaluated within a classic RCT model. The analysis will determine the effect of treatment on the primary outcome, change in Urogenital Distress Inventory (UDI) score at 6 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Botox A® injection (Active Comparator): A dose of 100 units of Botulinum toxin A will be injected into the bladder. Follow up visits at 2 weeks, 3 and 6 months post intervention to collect clinical and patient-reported outcomes.
  Interventions: Drug: Botox® injection
- Mid-urethral sling (Active Comparator): Mid-urethral Sling Procedure includes retropubic as well as transobturator full length slings. Follow up visits at 2 weeks, 3 and 6 months post intervention to collect clinical and patient-reported outcomes.
  Interventions: Device: Mid-urethral sling

INTERVENTIONS:
Drug: Botox® injection — Botulinum toxin A will be prepared by dissolving 100 units of botulinum toxin A into 10 ml of injectable saline. Indigo carmine or methylene blue 0.1 ml will be added to each syringe of botulinum toxin A. The treating physician will inject a total of 10 ml of the Botox A® into approximately 15 to 20 different detrusor muscle sites under direct visualization.
  Arms: Botox A® injection
Device: Mid-urethral sling — Mid-urethral Sling Procedure includes retropubic as well as transobturator full length slings. "Mini-sling" and "single-incision" sling will not be allowed due to potential risk for higher failure rate.
  Arms: Mid-urethral sling

SUMMARY:
The primary aim is to compare the effectiveness of intradetrusor injection of 100 unit injection of Botulinum toxin A to mid-urethral sling for change in MUI symptoms 6 months following treatment.

DETAILED DESCRIPTION:
Mixed urinary incontinence (MUI), defined as the presence of both stress urinary incontinence (SUI) and urgency urinary incontinence (UUI), is a challenging condition for which clinicians frequently use multiple sequential treatments that have undergone limited evaluation in rigorous clinical trials. The Mixed Urinary Incontinence: Mid-urethral Sling vs. Botox A (MUSA) trial will estimate the effect of Botulinum toxin A (Botox A ®) compared to mid-urethral sling for the treatment of MUI symptoms in 146 women. MUSA is a randomized 2-arm clinical trial.

The purpose of MUSA is to:

* compare treatment with either Botulinum toxin A (Botox A ®) or mid-urethral sling for women with MUI
* characterize patient characteristics associated with treatment response

The primary objective is to estimate the effect of intradetrusor injections Botulinum toxin A (Botox A ®) compared to mid-urethral sling for treatment of MUI in 146 women 6 months after treatment. The change in severity of MUI symptoms will be measured using the Urogenital Distress Inventory.

Secondary outcomes include:

• Urogenital Distress Inventory Stress and Irritative subscales

Other outcomes include:

* Urogenital Distress Inventory Obstructive subscale
* Patient bladder diary metrics including numbers of daily incontinence episodes and voids and voiding frequency
* Other patient reported outcomes/validated instruments and associated scales and subscales: EQ-5D, IIQ-LF, OABq-LF, OAB-SATq, PISQ-IR, PGI-I, PGI-S, PGSC, and SF-36
* Physical measures of effectiveness: Postvoid Residual Volume

The study will continue with an additional 6 month observational period until 12 months post treatment.

A supplemental study will characterize baseline putative proteins/protein pathways in women with MUI associated with change in UDI after treatment with MUS or onabotulinum toxin A. Those results are not reported with this record.

ELIGIBILITY:
Inclusion Criteria:

1. Reporting at least "moderate bother" from UUI item on UDI

   * "Do you experience urine leakage associated with a feeling of urgency?"
2. Reporting at least "moderate bother" from SUI item on UDI

   * "Do you experience urine leakage related to physical activity, coughing, or sneezing?"
3. Diagnosis of SUI defined by a positive cough stress test (CST) or UDE within the past 18 months
4. Presence of UUI on bladder diary with > 4 Urgency IE/3-day diary
5. Urinary symptoms >3 months
6. Persistent symptoms despite at least one or more conservative treatments (e.g. supervised behavioral therapy, physical therapy) as determined adequate by the physician.
7. Inadequate response to oral overactive bladder medications (including anti-cholinergic and/or beta-mimetic medication) unless patient is

   1. intolerant of oral overactive bladder medications, or
   2. oral overactive bladder medications are contraindicated as determined by the treating provider.
8. Urodynamics within past 18 months
9. Demonstrates ability (or have caregiver demonstrate ability) to perform clean intermittent self-catheterization.

Exclusion Criteria:

1. Anterior or apical compartment prolapse at or beyond the hymen (>0 on POPQ), regardless if patient is symptomatic

   * Women with anterior or apical prolapse above the hymen (<0) who do not report vaginal bulge symptoms will be eligible
2. Planned concomitant surgery for anterior vaginal wall or apical prolapse > 0

   * Women undergoing only rectocele repair or other repair unrelated to anterior or apical compartment are eligible
3. Women undergoing hysterectomy for any indication will be excluded
4. Active pelvic organ malignancy
5. Age <21 years
6. Pregnant or plans for future pregnancy in next 6 months, or within 12 months post-partum
7. Post-void residual >150 cc on 2 occasions within the past 6 months, or current catheter use
8. Participation in other trial that may influence results of this study
9. Unevaluated hematuria
10. Prior sling, synthetic mesh for prolapse, implanted nerve stimulator for urinary incontinence
11. Spinal cord injury or advanced/severe neurologic conditions including Multiple Sclerosis, Parkinsons, Myasthenia Gravis, Charcot-Marie-Tooth
12. Women on overactive bladder medication/therapy will be eligible after 3 week wash-out period
13. Non-ambulatory
14. History of serious adverse reaction to synthetic mesh
15. Not able to complete study assessments per clinician judgment, or not available for 6 month follow-up
16. Diagnosis of and/or history of bladder pain or chronic pelvic pain
17. Women who had intravesical Botox injection within the past 12 months
18. Women who have undergone anterior or apical pelvic organ prolapse repair within the past 6 months

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 150 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2024-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heidi S Harvey, MD, Principal Investigator — University of Pennsylvania; Marie Gantz, PhD, Principal Investigator — RTI International
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Department of Obstetrics and Gynecology, Birmingham, Alabama
  - University of California at San Diego, La Jolla, California
  - Kaiser Permanente, San Diego, California
  - Duke University, Duke Division of Urogynecology and Reconstructive Pelvic Surgery, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Magee-Women's Hospital, Department of Obstetrics and Gynecology, Pittsburgh, Pennsylvania
  - Brown/ Women and Infants Hospital of Rhode Island, Center for Women's Pelvic Medicine and Reconstructive Surgery, Providence, Rhode Island
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Harvie HS, Menefee SA, Richter HE, Sung VW, Chermansky CJ, Rahn DD, Amundsen CL, Arya LA, Rhodes E, Mazloomdoost D, Thomas S; National Institute of Child Health and Human Development Pelvic Floor Disorders Network. Midurethral Sling vs OnabotulinumtoxinA in Females With Urinary Incontinence: The MUSA Randomized Clinical Trial. JAMA. 2025 Jun 3;333(21):1887-1896. doi: 10.1001/jama.2025.4682. PMID 40323617
- [Derived] Harvie HS, Richter HE, Sung VW, Chermansky CJ, Menefee SA, Rahn DD, Amundsen CL, Arya LA, Huitema C, Mazloomdoost D, Thomas S; NICHD Pelvic Floor Disorders Network. Trial Design for Mixed Urinary Incontinence: Midurethral Sling Versus Botulinum Toxin A. Urogynecology (Phila). 2024 May 1;30(5):478-488. doi: 10.1097/SPV.0000000000001422. Epub 2024 Jan 11. PMID 38212101
- [Derived] Harvie HS, Sung VW, Neuwahl SJ, Honeycutt AA, Meyer I, Chermansky CJ, Menefee S, Hendrickson WK, Dunivan GC, Mazloomdoost D, Bass SJ, Gantz MG; Eunice Kennedy Shriver National Institute of Child Health and Human Development Pelvic Floor Disorders Network. Cost-effectiveness of behavioral and pelvic floor muscle therapy combined with midurethral sling surgery vs surgery alone among women with mixed urinary incontinence: results of the Effects of Surgical Treatment Enhanced With Exercise for Mixed Urinary Incontinence randomized trial. Am J Obstet Gynecol. 2021 Dec;225(6):651.e1-651.e26. doi: 10.1016/j.ajog.2021.06.099. Epub 2021 Jul 6. PMID 34242627

RESULTS

PARTICIPANT FLOW:
Groups:
- Botox A: Up to 2 administrations of Botulinum Toxin A
- Mid-Urethral Sling: Mid-Urethral Sling for treatment of urinary incontinence
Period: Overall Study
Arm/Group | Botox A | Mid-Urethral Sling
Started | 72 | 78
Received Treatment | 71 | 69
Provided Follow-up Data | 71 | 66
Completed | 66 | 63
Not Completed | 6 | 15
Not completed — Lost to Follow-up | 4 | 5
Not completed — Consent only through 6 months | 1 | 1
Not completed — Insurance did not cover procedure | 0 | 1
Not completed — Physician Decision | 0 | 3
Not completed — Withdrawal by Subject | 1 | 5

BASELINE CHARACTERISTICS:
Population: Baseline analysis is limited to those participants that were randomized, received treatment, and provided at least one post-baseline measurement.
Groups:
- Mid-Urethral Sling: Mid-Urethral Sling for treatment of urinary incont
- Total: Total of all reporting groups
Arm/Group | Botox A | Mid-Urethral Sling | Total
Number analyzed (Participants) | 71 | 66 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (11.4) | 59 (11.7) | 59 (11.5)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 71 | 66 | 137
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 0 | 2
  Black/African American | 10 | 10 | 20
  Native Hawaiian/Other Pacific Islander | 1 | 1 | 2
  Other | 3 | 1 | 4
  White | 55 | 54 | 109
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latina | 15 | 6 | 21
  Not Hispanic/Not Latina | 56 | 59 | 115
  Unknown/Not Reported | 0 | 1 | 1
Menopausal Status, Customized [Count of Participants; unit: Participants]
  Not sure | 8 | 3 | 11
  Post-menopausal | 56 | 49 | 105
  Pre-menopausal | 7 | 14 | 21
Education [Count of Participants; unit: Participants]
  4-Year College Degree | 21 | 11 | 32
  Associate College Degree | 17 | 13 | 30
  Graduate Degree | 8 | 8 | 16
  High School/GED | 19 | 29 | 48
  Less than High School | 3 | 2 | 5
  Unknown/Not Reported | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: UDI-LF Total Score Change From Baseline
Description: The Urogenital Distress Inventory is a standardized a measure of overactive bladder symptoms and health-related quality of life. The UDI scale has a range from 0 to 300 with higher scores indicating greater distress. The outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, 9, and 12 Months
Population: An intent-to-treat (ITT) analysis which included all eligible participants who were randomized and who provided outcome data after baseline was performed. Data that was collected after a participant was retreated for urinary incontinence was excluded from the analysis.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
units on a scale
  3.0: number analyzed (Participants) | 68 | 64
  3.0 | -82.2 [-100 to -64.4] | -84.6 [-101 to -68.3]
  6.0: number analyzed (Participants) | 64 | 65
  6.0 | -74.9 [-93.6 to -56.1] | -89.1 [-104.7 to -73.5]
  9.0: number analyzed (Participants) | 56 | 56
  9.0 | -63.1 [-81.8 to -44.5] | -85.6 [-102.7 to -68.6]
  12.0: number analyzed (Participants) | 61 | 60
  12.0 | -67.7 [-85.7 to -49.8] | -89.2 [-107.5 to -70.9]

2. Secondary Outcome: UDI-LF Stress Score Change From Baseline
Description: The Urogenital Distress Inventory is a standardized a measure of overactive bladder symptoms and health-related quality of life. The UDI Stress subscale has a range from 0 to 100 with higher scores indicating greater distress. The outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, 9, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
units on a scale
  3.0: number analyzed (Participants) | 68 | 64
  3.0 | -27.9 [-37.7 to -18.1] | -46.4 [-55.4 to -37.3]
  6.0: number analyzed (Participants) | 64 | 65
  6.0 | -30.2 [-39.6 to -20.9] | -45.1 [-53.6 to -36.7]
  9.0: number analyzed (Participants) | 56 | 56
  9.0 | -20.2 [-30.1 to -10.4] | -42.3 [-53.1 to -31.4]
  12.0: number analyzed (Participants) | 61 | 60
  12.0 | -24.3 [-34.6 to -14.1] | -44.4 [-53.8 to -35.1]

3. Secondary Outcome: UDI-LF Irritative Score Change From Baseline
Description: The Urogenital Distress Inventory is a standardized a measure of overactive bladder symptoms and health-related quality of life. The UDI Irritative subscale has a range from 0 to 100 with higher scores indicating greater distress. The outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, 9, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
units on a scale
  3.0: number analyzed (Participants) | 68 | 64
  3.0 | -40.8 [-47.3 to -34.2] | -28.1 [-35.6 to -20.6]
  6.0: number analyzed (Participants) | 64 | 65
  6.0 | -35.8 [-43.3 to -28.3] | -30.6 [-37.4 to -23.8]
  9.0: number analyzed (Participants) | 56 | 56
  9.0 | -32.7 [-40.5 to -25] | -30.8 [-38.8 to -22.7]
  12.0: number analyzed (Participants) | 61 | 60
  12.0 | -31.6 [-39 to -24.2] | -33 [-41.4 to -24.6]

4. Other Pre Specified Outcome: UDI-LF Obstructive Score Change From Baseline
Description: The Urogenital Distress Inventory is a standardized a measure of overactive bladder symptoms and health-related quality of life. The UDI Obstructive subscale has a range from 0 to 100 with higher scores indicating greater distress. The outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, 9, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
units on a scale
  3.0: number analyzed (Participants) | 68 | 64
  3.0 | -13.5 [-18.8 to -8.1] | -10.1 [-14.6 to -5.7]
  6.0: number analyzed (Participants) | 64 | 65
  6.0 | -8.9 [-13.8 to -4] | -13.4 [-17.5 to -9.3]
  9.0: number analyzed (Participants) | 56 | 56
  9.0 | -10.2 [-15.7 to -4.7] | -12.6 [-17 to -8.2]
  12.0: number analyzed (Participants) | 61 | 60
  12.0 | -11.8 [-16.4 to -7.2] | -11.7 [-16.5 to -6.9]

5. Other Pre Specified Outcome: Average Daily Frequency of Combined Mixed Stress/Urge and Non-categorized Incontinence Epsiodes Change From Baseline
Description: Based on data collected from participant-completed diaries, average daily frequency of combined mixed stress/urge and non-categorized incontinence epsiodes. The outcome variable is computed as the difference in number of episodes at 3, 6, and 12 months and the number of episodes at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: incontinence episodes/day
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 65 | 65
incontinence episodes/day
  3.0: number analyzed (Participants) | 59 | 61
  3.0 | -0.4 [-0.90 to 0.00] | -0.4 [-0.90 to 0.10]
  6.0: number analyzed (Participants) | 53 | 60
  6.0 | -0.2 [-0.50 to 0.10] | -0.7 [-1.10 to -0.30]
  12.0: number analyzed (Participants) | 53 | 56
  12.0 | -0.2 [-0.60 to 0.20] | -0.7 [-1.30 to -0.20]

6. Other Pre Specified Outcome: Average Daily Frequency of All Incontinence Epsiodes Change From Baseline
Description: Based on data collected from participant-completed diaries, average daily frequency of all incontinence epsiodes. The outcome variable is computed as the difference in number of episodes at 3, 6, and 12 months and the number of episodes at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: incontinence episodes/day
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 67 | 65
incontinence episodes/day
  3.0: number analyzed (Participants) | 61 | 61
  3.0 | -4 [-4.90 to -3.20] | -3.9 [-5.00 to -2.80]
  6.0: number analyzed (Participants) | 53 | 60
  6.0 | -3.2 [-3.90 to -2.40] | -4.1 [-5.20 to -3.10]
  12.0: number analyzed (Participants) | 53 | 56
  12.0 | -3.6 [-4.70 to -2.60] | -4.5 [-5.80 to -3.20]

7. Other Pre Specified Outcome: Average Daily Frequency of Diurnal Voids Change From Baseline
Description: Based on data collected from participant-completed diaries, average daily frequency of diurnal voids. The outcome variable is computed as the difference in number of voids at 3, 6, and 12 months and the number of voids at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: diurnal voids/day
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 67 | 65
diurnal voids/day
  3.0: number analyzed (Participants) | 61 | 61
  3.0 | -1.2 [-1.70 to -0.70] | 0 [-0.60 to 0.60]
  6.0: number analyzed (Participants) | 53 | 60
  6.0 | -0.8 [-1.30 to -0.20] | -0.2 [-0.90 to 0.60]
  12.0: number analyzed (Participants) | 53 | 56
  12.0 | -0.8 [-1.50 to -0.20] | -0.3 [-1.00 to 0.40]

8. Other Pre Specified Outcome: Average Daily Frequency of Nocturnal Voids Change From Baseline
Description: Based on data collected from participant-completed diaries, average daily frequency of nocturnal voids. The outcome variable is computed as the difference in number of voids at 3, 6, and 12 months and the number of voids at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: nocturnal voids/day
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 66 | 65
nocturnal voids/day
  3.0: number analyzed (Participants) | 60 | 61
  3.0 | -0.5 [-0.70 to -0.20] | -0.5 [-0.80 to -0.10]
  6.0: number analyzed (Participants) | 53 | 60
  6.0 | -0.3 [-0.60 to -0.10] | -0.2 [-0.50 to 0.20]
  12.0: number analyzed (Participants) | 53 | 56
  12.0 | -0.4 [-0.70 to -0.10] | -0.4 [-0.90 to 0.00]

9. Other Pre Specified Outcome: Average Daily Frequency of All Voids Change From Baseline
Description: Based on data collected from participant-completed diaries, average daily frequency of all voids. The outcome variable is computed as the difference in number of voids at 3, 6, and 12 months and the number of voids at baseline.
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: voids/day
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 67 | 65
voids/day
  3.0: number analyzed (Participants) | 61 | 61
  3.0 | -1.6 [-2.20 to -1.00] | -0.4 [-1.10 to 0.20]
  6.0: number analyzed (Participants) | 53 | 60
  6.0 | -1.1 [-1.70 to -0.50] | -0.4 [-1.10 to 0.40]
  12.0: number analyzed (Participants) | 53 | 56
  12.0 | -1.2 [-2.00 to -0.50] | -0.7 [-1.60 to 0.10]

10. Other Pre Specified Outcome: Normalization of Voiding Frequency
Description: Based on data collected from participant-completed diaries at baseline and 3, 6, and 12 months, for participants with >8 voids at baseline, the outcome is calculated as Yes=no more than 8 voids noted at the time point, No=Otherwise
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 43 | 40
Participants
  3.0: number analyzed (Participants) | 40 | 37
  3.0: No | 17 | 24
  3.0: Yes | 23 | 13
  6.0: number analyzed (Participants) | 35 | 35
  6.0: No | 17 | 25
  6.0: Yes | 18 | 10
  12.0: number analyzed (Participants) | 37 | 33
  12.0: No | 13 | 21
  12.0: Yes | 24 | 12

11. Other Pre Specified Outcome: Improvement of 50% or More in Voiding Frequency Post Baseline
Description: Based on data collected from participant-completed diaries at baseline and 3, 6, and 12 months, the outcome is calculated as Yes=at least 50% reduction in the number of voids between the timepoint and baseline, No=Otherwise
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 67 | 65
Participants
  3.0: number analyzed (Participants) | 61 | 61
  3.0: No | 60 | 61
  3.0: Yes | 1 | 0
  6.0: number analyzed (Participants) | 53 | 60
  6.0: No | 53 | 59
  6.0: Yes | 0 | 1
  12.0: number analyzed (Participants) | 53 | 56
  12.0: No | 50 | 54
  12.0: Yes | 3 | 2

12. Other Pre Specified Outcome: Worsening Voiding Frequency Post Baseline
Description: Based on data collected from participant-completed diaries at baseline and 3, 6, and 12 months, the outcome is calculated as Yes=greater than baseline number of voids at the time point or with greater than 8 voids at the time point, No=Otherwise
Time Frame: 3, 6, and 12 Months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 67 | 65
Participants
  3.0: number analyzed (Participants) | 61 | 61
  3.0: No | 49 | 39
  3.0: Yes | 12 | 22
  6.0: number analyzed (Participants) | 53 | 60
  6.0: No | 36 | 32
  6.0: Yes | 17 | 28
  12.0: number analyzed (Participants) | 53 | 56
  12.0: No | 37 | 34
  12.0: Yes | 16 | 22

13. Other Pre Specified Outcome: Change From Baseline EQ-5D Visual Analog Score
Description: EQ-5D is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life. The visual analog scale (VAS) score ranges from 0 to 100 with higher scores indicating a better quality of life. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 0.5 Months (2 Weeks) and 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 68 | 64
units on a scale
  0.5: number analyzed (Participants) | 62 | 62
  0.5 | 3.1 [-0.6 to 6.8] | 9.3 [4.7 to 13.8]
  3.0: number analyzed (Participants) | 61 | 57
  3.0 | 2.2 [-2.1 to 6.5] | 6.7 [1.9 to 11.5]
  6.0: number analyzed (Participants) | 60 | 62
  6.0 | 1.5 [-2.9 to 5.9] | 7.1 [3 to 11.3]
  9.0: number analyzed (Participants) | 52 | 53
  9.0 | 1.4 [-3.6 to 6.4] | 6.9 [2.8 to 11.1]
  12.0: number analyzed (Participants) | 56 | 53
  12.0 | 1.6 [-2.7 to 5.8] | 7.4 [2.3 to 12.5]

14. Other Pre Specified Outcome: Change From Baseline EQ-5D Index Score
Description: EQ-5D is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life. The index score ranges from 0 to 1 with higher scores indicating a better quality of life. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 0.5 Months (2 Weeks) and 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 70 | 64
units on a scale
  0.5: number analyzed (Participants) | 68 | 63
  0.5 | 0 [0 to 0] | 0 [0 to 0]
  3.0: number analyzed (Participants) | 65 | 60
  3.0 | 0 [0 to 0.1] | 0 [0 to 0.1]
  6.0: number analyzed (Participants) | 63 | 63
  6.0 | 0 [0 to 0.1] | 0 [0 to 0.1]
  9.0: number analyzed (Participants) | 53 | 52
  9.0 | 0 [-0.1 to 0] | 0 [0 to 0.1]
  12.0: number analyzed (Participants) | 58 | 54
  12.0 | 0 [0 to 0.1] | 0 [0 to 0.1]

15. Other Pre Specified Outcome: Change From Baseline IIQ-LF Physical Activity Score
Description: The Incontinence Impact Questionnaire-Long Form is a standardized a measure of health-related quality of life. The IIq-LF Physical Activity score ranges from 0 to 100 with higher scores indicating worse impact. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, 9, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
units on a scale
  3.0: number analyzed (Participants) | 67 | 64
  3.0 | -19.5 [-27.1 to -12] | -20.3 [-28 to -12.6]
  6.0: number analyzed (Participants) | 64 | 64
  6.0 | -20.7 [-26.2 to -15.2] | -21.1 [-28.5 to -13.8]
  9.0: number analyzed (Participants) | 55 | 56
  9.0 | -16.9 [-23.2 to -10.6] | -21.2 [-29 to -13.4]
  12.0: number analyzed (Participants) | 61 | 60
  12.0 | -18.1 [-24.5 to -11.7] | -25.3 [-32.9 to -17.8]

16. Other Pre Specified Outcome: Change From Baseline IIQ-LF Travel Score
Description: The Incontinence Impact Questionnaire-Long Form is a standardized a measure of health-related quality of life. The IIq-LF Travel score ranges from 0 to 100 with higher scores indicating worse impact. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, 9, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
units on a scale
  3.0: number analyzed (Participants) | 67 | 64
  3.0 | -19.6 [-27.6 to -11.7] | -22.2 [-30.5 to -13.9]
  6.0: number analyzed (Participants) | 64 | 64
  6.0 | -23.3 [-29.4 to -17.1] | -25.4 [-33.7 to -17.1]
  9.0: number analyzed (Participants) | 55 | 56
  9.0 | -14.3 [-21 to -7.7] | -25.8 [-34.5 to -17]
  12.0: number analyzed (Participants) | 61 | 60
  12.0 | -19.7 [-26.2 to -13.3] | -28.1 [-36.7 to -19.6]

17. Other Pre Specified Outcome: Change From Baseline IIQ-LF Social/Relationships Score
Description: The Incontinence Impact Questionnaire-Long Form is a standardized a measure of health-related quality of life. The IIq-LF Social Relationship score ranges from 0 to 100 with higher scores indicating worse impact. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, 9, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
units on a scale
  3.0: number analyzed (Participants) | 67 | 64
  3.0 | -15.7 [-22.6 to -8.7] | -18.9 [-26.8 to -11]
  6.0: number analyzed (Participants) | 64 | 64
  6.0 | -16.9 [-22.8 to -11] | -20.3 [-27.8 to -12.8]
  9.0: number analyzed (Participants) | 55 | 56
  9.0 | -10.3 [-15.8 to -4.7] | -19.9 [-27.8 to -12]
  12.0: number analyzed (Participants) | 61 | 60
  12.0 | -15.7 [-21.8 to -9.5] | -22.3 [-30.7 to -13.9]

18. Other Pre Specified Outcome: Change From Baseline IIQ-LF Emotional Health Score
Description: The Incontinence Impact Questionnaire-Long Form is a standardized a measure of health-related quality of life. The IIq-LF Emotional Health score ranges from 0 to 100 with higher scores indicating worse impact. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, 9, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
units on a scale
  3.0: number analyzed (Participants) | 68 | 64
  3.0 | -17.7 [-24.8 to -10.6] | -19.5 [-26 to -12.9]
  6.0: number analyzed (Participants) | 64 | 64
  6.0 | -20.2 [-26.5 to -13.9] | -21.5 [-28.3 to -14.8]
  9.0: number analyzed (Participants) | 55 | 56
  9.0 | -12.5 [-19.4 to -5.6] | -19.7 [-26 to -13.5]
  12.0: number analyzed (Participants) | 61 | 60
  12.0 | -17.5 [-24.5 to -10.5] | -26.8 [-35.2 to -18.4]

19. Other Pre Specified Outcome: Change From Baseline IIQ-LF Total Score
Description: The Incontinence Impact Questionnaire-Long Form is a standardized a measure of health-related quality of life. The IIq-LF Total score ranges from 0 to 400 with higher scores indicating worse impact. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, 9, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
units on a scale
  3.0: number analyzed (Participants) | 67 | 64
  3.0 | -72.9 [-99.5 to -46.2] | -80.8 [-108.4 to -53.2]
  6.0: number analyzed (Participants) | 64 | 64
  6.0 | -81.1 [-101.3 to -60.9] | -88.4 [-115.4 to -61.4]
  9.0: number analyzed (Participants) | 55 | 56
  9.0 | -54 [-75.7 to -32.2] | -86.6 [-113.9 to -59.3]
  12.0: number analyzed (Participants) | 61 | 60
  12.0 | -71 [-93.4 to -48.6] | -102.5 [-133.1 to -71.9]

20. Other Pre Specified Outcome: Change From Baseline OABq-LF Symptom Severity Score
Description: The Overactive Bladder Questionnaire-Long Form is a standardized a measure of overactive bladder symptoms and health-related quality of life. The OABq-LF Symptom Severity score ranges from 0 to 100 with higher score indicating worse quality of life. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, 9, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
units on a scale
  3.0: number analyzed (Participants) | 68 | 64
  3.0 | -41 [-47.9 to -34] | -28.7 [-36.6 to -20.7]
  6.0: number analyzed (Participants) | 64 | 65
  6.0 | -34.3 [-41 to -27.6] | -32 [-39.6 to -24.3]
  9.0: number analyzed (Participants) | 55 | 56
  9.0 | -26.7 [-33.9 to -19.4] | -28.8 [-37.5 to -20.1]
  12.0: number analyzed (Participants) | 61 | 60
  12.0 | -30.6 [-38.3 to -22.8] | -36.1 [-44.3 to -27.9]

21. Other Pre Specified Outcome: Change From Baseline OABq-LF Coping Score
Description: The Overactive Bladder Questionnaire-Long Form is a standardized a measure of overactive bladder symptoms and health-related quality of life. The OABq-LF Coping score ranges from 0 to 100 with higher score indicating better quality of life. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, 9, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
units on a scale
  3.0: number analyzed (Participants) | 67 | 64
  3.0 | 29.7 [21.7 to 37.8] | 29.5 [21.9 to 37.1]
  6.0: number analyzed (Participants) | 64 | 65
  6.0 | 24.3 [17.2 to 31.4] | 29.8 [22 to 37.5]
  9.0: number analyzed (Participants) | 55 | 56
  9.0 | 18.8 [11.8 to 25.8] | 26.4 [18 to 34.9]
  12.0: number analyzed (Participants) | 61 | 60
  12.0 | 24.7 [17.9 to 31.5] | 34.4 [25.6 to 43.2]

22. Other Pre Specified Outcome: Change From Baseline OABq-LF Concern Score
Description: The Overactive Bladder Questionnaire-Long Form is a standardized a measure of overactive bladder symptoms and health-related quality of life. The OABq-LF Concern score ranges from 0 to 100 with higher score indicating better quality of life. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, 9, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
units on a scale
  3.0: number analyzed (Participants) | 67 | 64
  3.0 | 32.3 [24.6 to 40] | 29.6 [22.3 to 36.9]
  6.0: number analyzed (Participants) | 64 | 65
  6.0 | 26.1 [19.7 to 32.5] | 31.2 [23.7 to 38.7]
  9.0: number analyzed (Participants) | 55 | 56
  9.0 | 16.7 [9.2 to 24.2] | 28.2 [20.3 to 36.1]
  12.0: number analyzed (Participants) | 61 | 60
  12.0 | 24.5 [16.8 to 32.2] | 35.6 [27.1 to 44.1]

23. Other Pre Specified Outcome: Change From Baseline OABq-LF Sleep Score
Description: The Overactive Bladder Questionnaire-Long Form is a standardized a measure of overactive bladder symptoms and health-related quality of life. The OABq-LF Sleep score ranges from 0 to 100 with higher score indicating better quality of life. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, 9, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
units on a scale
  3.0: number analyzed (Participants) | 67 | 64
  3.0 | 23.8 [16.3 to 31.3] | 20.7 [12.4 to 29]
  6.0: number analyzed (Participants) | 64 | 65
  6.0 | 21.6 [14.4 to 28.8] | 18.4 [10.8 to 25.9]
  9.0: number analyzed (Participants) | 55 | 56
  9.0 | 15.6 [8.4 to 22.7] | 19 [11.4 to 26.7]
  12.0: number analyzed (Participants) | 61 | 60
  12.0 | 16.8 [9.3 to 24.3] | 19.8 [9.7 to 29.8]

24. Other Pre Specified Outcome: Change From Baseline OABq-LF Social Score
Description: The Overactive Bladder Questionnaire-Long Form is a standardized a measure of overactive bladder symptoms and health-related quality of life. The OABq-LF Social score ranges from 0 to 100 with higher score indicating better quality of life. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, 9, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
units on a scale
  3.0: number analyzed (Participants) | 68 | 64
  3.0 | 15.1 [8.7 to 21.5] | 20 [13 to 27]
  6.0: number analyzed (Participants) | 64 | 65
  6.0 | 11.8 [5.5 to 18] | 19.6 [13.4 to 25.8]
  9.0: number analyzed (Participants) | 55 | 56
  9.0 | 4.8 [-0.5 to 10.1] | 18.4 [10.9 to 26]
  12.0: number analyzed (Participants) | 61 | 60
  12.0 | 11 [4.7 to 17.4] | 21 [13.6 to 28.4]

25. Other Pre Specified Outcome: Change From Baseline OABq-LF HRQL Total Score
Description: The Overactive Bladder Questionnaire-Long Form is a standardized a measure of overactive bladder symptoms and health-related quality of life. The OABq-LF HRQL score ranges from 0 to 100 with higher score indicating better quality of life. The change from baseline outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 3, 6, 9, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
units on a scale
  3.0: number analyzed (Participants) | 67 | 64
  3.0 | 26.4 [19.8 to 33] | 25.9 [19.2 to 32.6]
  6.0: number analyzed (Participants) | 64 | 65
  6.0 | 21.8 [16 to 27.5] | 25.9 [19.4 to 32.3]
  9.0: number analyzed (Participants) | 55 | 56
  9.0 | 14.8 [9.2 to 20.4] | 23.9 [16.8 to 30.9]
  12.0: number analyzed (Participants) | 61 | 60
  12.0 | 20.3 [14.3 to 26.4] | 29.1 [21.4 to 36.9]

26. Other Pre Specified Outcome: OAB-SATq-LF Satisfaction Score
Description: The Overactive Bladder Satisfaction with Treatment Questionnaire is a standardized a measure of satisfaction with treatment for overactive bladder symptoms. The OAB-SATq Satisfaction score ranges from 0 to 100 with higher scores indicating higher satisfaction.
Time Frame: 3, 6, 9, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
units on a scale
  3.0: number analyzed (Participants) | 68 | 62
  3.0 | 65.7 [58.7 to 72.7] | 60.1 [51.9 to 68.3]
  6.0: number analyzed (Participants) | 64 | 65
  6.0 | 64.5 [57.6 to 71.3] | 60.3 [52.5 to 68.2]
  9.0: number analyzed (Participants) | 55 | 56
  9.0 | 64.4 [57.5 to 71.2] | 57.5 [48.8 to 66.2]
  12.0: number analyzed (Participants) | 61 | 60
  12.0 | 60.4 [53 to 67.8] | 56.3 [46.8 to 65.9]

27. Other Pre Specified Outcome: OAB-SATq-LF Side Effects Score
Description: The Overactive Bladder Satisfaction with Treatment Questionnaire is a standardized a measure of satisfaction with treatment for overactive bladder symptoms. The OAB-SATq Side Effect score ranges from 0 to 100 with higher scores indicating fewer side effects.
Time Frame: 3, 6, 9, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
units on a scale
  3.0: number analyzed (Participants) | 67 | 64
  3.0 | 91.9 [87.5 to 96.4] | 93.5 [89.7 to 97.3]
  6.0: number analyzed (Participants) | 63 | 65
  6.0 | 89 [83.5 to 94.5] | 87.4 [81.5 to 93.4]
  9.0: number analyzed (Participants) | 55 | 56
  9.0 | 90.2 [84.4 to 95.9] | 86.3 [79.7 to 92.9]
  12.0: number analyzed (Participants) | 61 | 60
  12.0 | 91.8 [87 to 96.6] | 88.5 [82.2 to 94.8]

28. Other Pre Specified Outcome: OAB-SATq-LF Endorsement Score
Description: The Overactive Bladder Satisfaction with Treatment Questionnaire is a standardized a measure of satisfaction with treatment for overactive bladder symptoms. The OAB-SATq Endorsement score ranges from 0 to 100 with higher scores indicating greater endorsement.
Time Frame: 3, 6, 9, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
units on a scale
  3.0: number analyzed (Participants) | 68 | 64
  3.0 | 74.3 [67.8 to 80.9] | 67.9 [59.8 to 76]
  6.0: number analyzed (Participants) | 64 | 65
  6.0 | 72 [64.4 to 79.6] | 68.3 [60.5 to 76]
  9.0: number analyzed (Participants) | 55 | 56
  9.0 | 77.7 [70.5 to 84.9] | 73.6 [65.6 to 81.7]
  12.0: number analyzed (Participants) | 61 | 60
  12.0 | 71.7 [63.8 to 79.5] | 68.2 [59 to 77.3]

29. Other Pre Specified Outcome: OAB-SATq-LF Convenience Score
Description: The Overactive Bladder Satisfaction with Treatment Questionnaire is a standardized a measure of satisfaction with treatment for overactive bladder symptoms. The OAB-SATq Convenience score ranges from 0 to 100 with higher scores indicating greater convenience.
Time Frame: 3, 6, 9, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
units on a scale
  3.0: number analyzed (Participants) | 67 | 64
  3.0 | 64.2 [57.6 to 70.7] | 64.1 [56.7 to 71.4]
  6.0: number analyzed (Participants) | 62 | 65
  6.0 | 66.5 [59.3 to 73.6] | 66.8 [60 to 73.5]
  9.0: number analyzed (Participants) | 55 | 55
  9.0 | 67.6 [62.5 to 72.8] | 64.7 [58.1 to 71.3]
  12.0: number analyzed (Participants) | 61 | 60
  12.0 | 65.6 [59.7 to 71.4] | 66.3 [58.5 to 74.2]

30. Other Pre Specified Outcome: OAB-SAT-q Preference Indicator
Description: The Overactive Bladder Satisfaction with Treatment Questionnaire is a standardized a measure of satisfaction with treatment for overactive bladder symptoms. The preference score is a binary [yes/no] indicator as to whether a subject indicated slight or definite preference for the treatment among women that have had previous treatment for overactive bladder. The outcome is the percentage of participants that prefer the current treatment to previous treatments.
Time Frame: 3, 6, 9, and 12 Months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
Participants
  3.0: number analyzed (Participants) | 68 | 64
  3.0: Unknown | 16 | 24
  3.0: No | 5 | 5
  3.0: Yes | 47 | 35
  6.0: number analyzed (Participants) | 64 | 65
  6.0: Unknown | 17 | 21
  6.0: No | 6 | 8
  6.0: Yes | 41 | 36
  9.0: number analyzed (Participants) | 55 | 56
  9.0: Unknown | 17 | 15
  9.0: No | 5 | 5
  9.0: Yes | 33 | 36
  12.0: number analyzed (Participants) | 61 | 60
  12.0: Unknown | 15 | 19
  12.0: No | 10 | 7
  12.0: Yes | 36 | 34

31. Other Pre Specified Outcome: PGI-I Score Binary Improvement Indicator
Description: The Patient Global Impression of Improvement (PGI-I) is a patient-reported measure of perceived improvement with treatment, as assessed on a scale of 1 (very much better) to 7 (very much worse). Included here are participants who had improvement as indicated by a rating of 1 (very much better), 2 (much better).
Time Frame: 3, 6, 9, and 12 Months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
Participants
  3.0: number analyzed (Participants) | 68 | 64
  3.0: No | 28 | 30
  3.0: Yes | 40 | 34
  6.0: number analyzed (Participants) | 64 | 65
  6.0: No | 25 | 33
  6.0: Yes | 39 | 32
  9.0: number analyzed (Participants) | 56 | 56
  9.0: No | 22 | 25
  9.0: Yes | 34 | 31
  12.0: number analyzed (Participants) | 61 | 60
  12.0: No | 35 | 31
  12.0: Yes | 26 | 29

32. Other Pre Specified Outcome: PGI-S Score Binary Condition Severity Indicator
Description: The Patient Global Impression of Severity (PGI-S) is a patient-reported measure of perceived severity of condition, as assessed on a scale of 1 (Normal) to 4 (Severe). Included here are participants who reported Normal or Mild severity as indicated by a rating of 1 or 2.
Time Frame: Baseline and 3, 6, 9, and 12 Months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
Participants
  Baseline: number analyzed (Participants) | 70 | 63
  Baseline: No | 57 | 53
  Baseline: Yes | 13 | 10
  3.0: number analyzed (Participants) | 68 | 64
  3.0: No | 29 | 30
  3.0: Yes | 39 | 34
  6.0: number analyzed (Participants) | 64 | 65
  6.0: No | 29 | 29
  6.0: Yes | 35 | 36
  9.0: number analyzed (Participants) | 56 | 56
  9.0: No | 27 | 24
  9.0: Yes | 29 | 32
  12.0: number analyzed (Participants) | 61 | 60
  12.0: No | 28 | 24
  12.0: Yes | 33 | 36

33. Other Pre Specified Outcome: PGSC Score Binary Improvement Indicator
Description: Patient GLobal Impression of Symptom Control(PGSC) is a patient-reported measure of perceived adequate symptom control, as assessed on a scale of 1 (disagree strongly) to 5 (agree strongly). Included here are participants who had adequate control as indicated by a rating of 5 (agree strongly) or 4 (agree).
Time Frame: 3, 6, 9, and 12 Months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
Participants
  3.0: number analyzed (Participants) | 68 | 64
  3.0: No | 32 | 28
  3.0: Yes | 36 | 36
  6.0: number analyzed (Participants) | 64 | 65
  6.0: No | 30 | 33
  6.0: Yes | 34 | 32
  9.0: number analyzed (Participants) | 56 | 56
  9.0: No | 28 | 27
  9.0: Yes | 28 | 29
  12.0: number analyzed (Participants) | 62 | 60
  12.0: No | 33 | 24
  12.0: Yes | 29 | 36

34. Other Pre Specified Outcome: Change From Baseline PISQ-IR NSA-PR Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised measures the impact of incontinence symptoms on sexual function and satisfaction. The Not Sexually Active-Partner Related (NSA-PR) ranges from 1 to 4 with higher scores indicating greater sexual function. The outcome is calculated as the difference in score at 3, 6, 9, and 12 months and the score at baseline.
Time Frame: 3, 6, 9, and 12 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 33 | 35
units on a scale
  3.0: number analyzed (Participants) | 29 | 32
  3.0 | 0.3 [-0.1 to 0.7] | 0.3 [0.1 to 0.5]
  6.0: number analyzed (Participants) | 26 | 32
  6.0 | 0 [-0.4 to 0.4] | 0.3 [0 to 0.6]
  9.0: number analyzed (Participants) | 21 | 24
  9.0 | 0.1 [-0.3 to 0.6] | 0.1 [-0.3 to 0.5]
  12.0: number analyzed (Participants) | 26 | 28
  12.0 | 0.3 [0 to 0.6] | 0.1 [-0.3 to 0.4]

35. Other Pre Specified Outcome: Change From Baseline PISQ-IR NSA-CS Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised measures the impact of incontinence symptoms on sexual function and satisfaction. The Not Sexually Active-Condition Specific (NSA-CS) ranges from 1 to 4 with higher scores indicating greater sexual function. The outcome is calculated as the difference in score at 3, 6, 9, and 12 months and the score at baseline.
Time Frame: 3, 6, 9, and 12 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 32 | 34
units on a scale
  3.0: number analyzed (Participants) | 25 | 29
  3.0 | -0.2 [-0.5 to 0] | -0.1 [-0.5 to 0.2]
  6.0: number analyzed (Participants) | 22 | 29
  6.0 | -0.2 [-0.7 to 0.2] | 0 [-0.3 to 0.4]
  9.0: number analyzed (Participants) | 19 | 22
  9.0 | -0.2 [-0.4 to 0.1] | -0.1 [-0.4 to 0.2]
  12.0: number analyzed (Participants) | 24 | 25
  12.0 | 0.2 [-0.1 to 0.6] | -0.3 [-0.7 to 0.2]

36. Other Pre Specified Outcome: Change From Baseline PISQ-IR NSA-GQA Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised measures the impact of incontinence symptoms on sexual function and satisfaction. The Not Sexually Active-Global Quality Rating (NSA-GQA) ranges from 1 to 4.5 with higher scores indicating greater sexual function. The outcome is calculated as the difference in score at 3, 6, 9, and 12 months and the score at baseline.
Time Frame: 3, 6, 9, and 12 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 32 | 34
units on a scale
  3.0: number analyzed (Participants) | 27 | 30
  3.0 | -0.1 [-0.5 to 0.2] | -0.3 [-0.6 to 0.1]
  6.0: number analyzed (Participants) | 23 | 32
  6.0 | -0.3 [-0.8 to 0.2] | -0.3 [-0.8 to 0.1]
  9.0: number analyzed (Participants) | 21 | 25
  9.0 | -0.2 [-0.8 to 0.4] | -0.4 [-0.8 to -0.1]
  12.0: number analyzed (Participants) | 25 | 27
  12.0 | -0.4 [-0.9 to 0.1] | -0.2 [-0.7 to 0.2]

37. Other Pre Specified Outcome: Change From Baseline PISQ-IR NSA-CI Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised measures the impact of incontinence symptoms on sexual function and satisfaction. The Not Sexually Active-Condition Impact (NSA-CI) ranges from 1 to 4 with higher scores indicating greater sexual function. The outcome is calculated as the difference in score at 3, 6, 9, and 12 months and the score at baseline.
Time Frame: 3, 6, 9, and 12 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 32 | 35
units on a scale
  3.0: number analyzed (Participants) | 27 | 31
  3.0 | -0.3 [-0.6 to 0] | -0.4 [-0.8 to 0]
  6.0: number analyzed (Participants) | 24 | 33
  6.0 | -0.3 [-0.7 to 0.1] | -0.3 [-0.8 to 0.1]
  9.0: number analyzed (Participants) | 21 | 25
  9.0 | -0.3 [-0.8 to 0.1] | -0.2 [-0.7 to 0.2]
  12.0: number analyzed (Participants) | 25 | 27
  12.0 | -0.2 [-0.5 to 0.1] | -0.4 [-0.8 to 0]

38. Other Pre Specified Outcome: Change From Baseline PISQ-IR SA-AO Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised measures the impact of incontinence symptoms on sexual function and satisfaction. The Sexually Active-Arousal Orgasm (SA-AO) ranges from 1 to 5 with higher scores indicating greater sexual function. The outcome is calculated as the difference in score at 3, 6, 9, and 12 months and the score at baseline.
Time Frame: 3, 6, 9, and 12 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 31 | 28
units on a scale
  3.0: number analyzed (Participants) | 28 | 22
  3.0 | 0 [-0.1 to 0.2] | -0.1 [-0.5 to 0.3]
  6.0: number analyzed (Participants) | 26 | 22
  6.0 | 0 [-0.2 to 0.2] | 0.1 [-0.2 to 0.3]
  9.0: number analyzed (Participants) | 23 | 20
  9.0 | -0.1 [-0.4 to 0.2] | 0.1 [-0.2 to 0.3]
  12.0: number analyzed (Participants) | 22 | 21
  12.0 | 0 [-0.3 to 0.3] | 0 [-0.3 to 0.2]

39. Other Pre Specified Outcome: Change From Baseline PISQ-IR SA-PR Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised measures the impact of incontinence symptoms on sexual function and satisfaction. The Sexually Active-Partner Related (SA-PR) ranges from 1 to 4 with higher scores indicating greater sexual function. The outcome is calculated as the difference in score at 3, 6, 9, and 12 months and the score at baseline.
Time Frame: 3, 6, 9, and 12 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 28 | 26
units on a scale
  3.0: number analyzed (Participants) | 26 | 21
  3.0 | 0 [-0.3 to 0.2] | 0 [-0.3 to 0.2]
  6.0: number analyzed (Participants) | 24 | 18
  6.0 | 0 [-0.2 to 0.3] | 0.1 [-0.2 to 0.5]
  9.0: number analyzed (Participants) | 22 | 18
  9.0 | -0.1 [-0.3 to 0.2] | -0.3 [-0.6 to 0]
  12.0: number analyzed (Participants) | 18 | 21
  12.0 | -0.1 [-0.5 to 0.2] | -0.1 [-0.4 to 0.1]

40. Other Pre Specified Outcome: Change From Baseline PISQ-IR SA-CS Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised measures the impact of incontinence symptoms on sexual function and satisfaction. The Sexually Active-Condition Specific (SA-CS) ranges from 1 to 5 with higher scores indicating greater sexual function. The outcome is calculated as the difference in score at 3, 6, 9, and 12 months and the score at baseline.
Time Frame: 3, 6, 9, and 12 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 30 | 25
units on a scale
  3.0: number analyzed (Participants) | 27 | 19
  3.0 | 0.5 [0.2 to 0.7] | 0.5 [0.1 to 0.8]
  6.0: number analyzed (Participants) | 24 | 20
  6.0 | 0.3 [0 to 0.6] | 0.6 [0.1 to 1]
  9.0: number analyzed (Participants) | 21 | 18
  9.0 | 0.3 [-0.1 to 0.6] | 0.2 [-0.4 to 0.8]
  12.0: number analyzed (Participants) | 21 | 18
  12.0 | 0.3 [-0.1 to 0.6] | 0.4 [-0.2 to 1.1]

41. Other Pre Specified Outcome: Change From Baseline PISQ-IR SA-GQR Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised measures the impact of incontinence symptoms on sexual function and satisfaction. The Sexually Active-Global Quality Rating (SA-GQR) ranges from 1 to 4.75 with higher scores indicating greater sexual function. The outcome is calculated as the difference in score at 3, 6, 9, and 12 months and the score at baseline.
Time Frame: 3, 6, 9, and 12 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 30 | 28
units on a scale
  3.0: number analyzed (Participants) | 27 | 22
  3.0 | 0 [-0.4 to 0.3] | 0.3 [-0.1 to 0.7]
  6.0: number analyzed (Participants) | 25 | 22
  6.0 | 0 [-0.3 to 0.4] | 0.2 [-0.2 to 0.5]
  9.0: number analyzed (Participants) | 22 | 20
  9.0 | -0.1 [-0.6 to 0.3] | -0.4 [-0.9 to 0.1]
  12.0: number analyzed (Participants) | 21 | 21
  12.0 | -0.1 [-0.4 to 0.3] | -0.2 [-0.5 to 0.2]

42. Other Pre Specified Outcome: Change From Baseline PISQ-IR SA-CI Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised measures the impact of incontinence symptoms on sexual function and satisfaction. The Sexually Active-Condition Impact (SA-CI) ranges from 1 to 4 with higher scores indicating greater sexual function. The outcome is calculated as the difference in score at 3, 6, 9, and 12 months and the score at baseline.
Time Frame: 3, 6, 9, and 12 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 31 | 28
units on a scale
  3.0: number analyzed (Participants) | 28 | 22
  3.0 | 0.4 [0.1 to 0.7] | 0.6 [0.3 to 1]
  6.0: number analyzed (Participants) | 25 | 22
  6.0 | 0.2 [-0.1 to 0.5] | 0.8 [0.4 to 1.1]
  9.0: number analyzed (Participants) | 23 | 20
  9.0 | 0.3 [0 to 0.6] | 0.3 [-0.1 to 0.7]
  12.0: number analyzed (Participants) | 22 | 21
  12.0 | 0.3 [-0.1 to 0.6] | 0.9 [0.5 to 1.4]

43. Other Pre Specified Outcome: Change From Baseline PISQ-IR SA-D Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised measures the impact of incontinence symptoms on sexual function and satisfaction. The Sexually Active-Desire (SA-D) ranges from 1 to 5 with higher scores indicating greater sexual function. The outcome is calculated as the difference in score at 3, 6, 9, and 12 months and the score at baseline.
Time Frame: 3, 6, 9, and 12 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 30 | 28
units on a scale
  3.0: number analyzed (Participants) | 27 | 22
  3.0 | 0.1 [-0.1 to 0.4] | 0.1 [-0.2 to 0.3]
  6.0: number analyzed (Participants) | 25 | 22
  6.0 | 0 [-0.2 to 0.1] | -0.1 [-0.3 to 0.1]
  9.0: number analyzed (Participants) | 23 | 20
  9.0 | 0 [-0.3 to 0.2] | 0.1 [-0.2 to 0.4]
  12.0: number analyzed (Participants) | 21 | 21
  12.0 | -0.2 [-0.5 to 0.1] | 0 [-0.3 to 0.4]

44. Other Pre Specified Outcome: Change From Baseline PISQ-IR SA Average Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised measures the impact of incontinence symptoms on sexual function and satisfaction. The Sexually Active-Average (SA-AVG) ranges from 1 to 5 with higher scores indicating greater sexual function. The outcome is calculated as the difference in score at 3, 6, 9, and 12 months and the score at baseline.
Time Frame: 3, 6, 9, and 12 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 31 | 28
units on a scale
  3.0: number analyzed (Participants) | 28 | 22
  3.0 | 0.2 [0 to 0.3] | 0.2 [0.1 to 0.4]
  6.0: number analyzed (Participants) | 26 | 22
  6.0 | 0.1 [-0.1 to 0.2] | 0.3 [0.1 to 0.5]
  9.0: number analyzed (Participants) | 23 | 20
  9.0 | 0 [-0.1 to 0.2] | 0 [-0.2 to 0.2]
  12.0: number analyzed (Participants) | 20 | 21
  12.0 | 0 [-0.2 to 0.2] | 0.2 [0 to 0.4]

45. Other Pre Specified Outcome: SF-36 Physical Functioning Score
Description: SF-36 is a standardized survey evaluating 8 domains of functional health and wellbeing: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for physical function domain was an average of the individual question scores of this domain, which are scaled 0-100 (100=highest level of functioning). The outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 0.5 Months (2 Weeks) and 3, 6, 9, and 12 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
units on a scale
  0.5: number analyzed (Participants) | 69 | 63
  0.5 | 12.9 [6.3 to 19.5] | 12.2 [6.3 to 18.1]
  3.0: number analyzed (Participants) | 68 | 64
  3.0 | 10.9 [4.8 to 17] | 13.9 [7.1 to 20.6]
  6.0: number analyzed (Participants) | 63 | 64
  6.0 | 10.5 [4.6 to 16.3] | 14 [7.1 to 20.9]
  9.0: number analyzed (Participants) | 55 | 56
  9.0 | 8.9 [1.8 to 15.9] | 9.7 [3.6 to 15.7]
  12.0: number analyzed (Participants) | 61 | 60
  12.0 | 10 [4.1 to 15.9] | 13.3 [6.5 to 20]

46. Other Pre Specified Outcome: SF-36 Role Physical Score
Description: SF-36 is a standardized survey evaluating 8 domains of functional health and wellbeing: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for physical role limitations domain was an average of the individual question scores of this domain, which are scaled 0-100 (100=highest level of functioning). The outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 0.5 Months (2 Weeks) and 3, 6, 9, and 12 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
units on a scale
  0.5: number analyzed (Participants) | 69 | 63
  0.5 | 14.1 [3.1 to 25.2] | -1.2 [-12.7 to 10.3]
  3.0: number analyzed (Participants) | 68 | 64
  3.0 | 12.5 [2.2 to 22.8] | 11.3 [1.6 to 21.1]
  6.0: number analyzed (Participants) | 63 | 64
  6.0 | 12.3 [1.7 to 22.9] | 12.1 [2 to 22.2]
  9.0: number analyzed (Participants) | 55 | 55
  9.0 | 3.6 [-8.3 to 15.6] | 7.7 [-4.3 to 19.8]
  12.0: number analyzed (Participants) | 61 | 60
  12.0 | 8.6 [-1.2 to 18.4] | 4.9 [-7.3 to 17.1]

47. Other Pre Specified Outcome: SF-36 Bodily Pain Score
Description: SF-36 is a standardized survey evaluating 8 domains of functional health and wellbeing: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for bodily pain domain was an average of the individual question scores of this domain, which are scaled 0-100 (100=highest level of functioning). The outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 0.5 Months (2 Weeks) and 3, 6, 9, and 12 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
units on a scale
  0.5: number analyzed (Participants) | 69 | 63
  0.5 | 2.6 [-3 to 8.2] | 2.4 [-3.6 to 8.5]
  3.0: number analyzed (Participants) | 68 | 64
  3.0 | 5.1 [-0.6 to 10.9] | 0.6 [-5.4 to 6.5]
  6.0: number analyzed (Participants) | 63 | 64
  6.0 | -0.4 [-6.3 to 5.5] | 0.8 [-5.1 to 6.6]
  9.0: number analyzed (Participants) | 55 | 56
  9.0 | -1.6 [-8.1 to 5] | 4.2 [-1.8 to 10.2]
  12.0: number analyzed (Participants) | 61 | 60
  12.0 | -0.8 [-6.9 to 5.2] | 6.4 [0.1 to 12.7]

48. Other Pre Specified Outcome: SF-36 General Health Score
Description: SF-36 is a standardized survey evaluating 8 domains of functional health and wellbeing: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for general health domain was an average of the individual question scores of this domain, which are scaled 0-100 (100=highest level of functioning). The outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 0.5 Months (2 Weeks) and 3, 6, 9, and 12 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
units on a scale
  0.5: number analyzed (Participants) | 69 | 63
  0.5 | 5.2 [1.9 to 8.4] | 2.5 [-1.2 to 6.3]
  3.0: number analyzed (Participants) | 68 | 64
  3.0 | 2.4 [-1.3 to 6] | -1.7 [-5.8 to 2.5]
  6.0: number analyzed (Participants) | 63 | 64
  6.0 | 2.6 [-1.4 to 6.7] | -0.6 [-4.4 to 3.2]
  9.0: number analyzed (Participants) | 55 | 56
  9.0 | -1.6 [-6 to 2.7] | -2.2 [-6.5 to 2.2]
  12.0: number analyzed (Participants) | 61 | 60
  12.0 | -1.1 [-5.3 to 3.1] | -0.3 [-4.8 to 4.1]

49. Other Pre Specified Outcome: SF-36 Vitality Score
Description: SF-36 is a standardized survey evaluating 8 domains of functional health and wellbeing: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for vitality domain was an average of the individual question scores of this domain, which are scaled 0-100 (100=highest level of functioning). The outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 0.5 Months (2 Weeks) and 3, 6, 9, and 12 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
units on a scale
  0.5: number analyzed (Participants) | 69 | 63
  0.5 | 6.1 [1 to 11.1] | 6.5 [1.8 to 11.3]
  3.0: number analyzed (Participants) | 68 | 64
  3.0 | 3.5 [-1.7 to 8.6] | 5.3 [0.6 to 10.1]
  6.0: number analyzed (Participants) | 63 | 64
  6.0 | 4.7 [-0.1 to 9.5] | 3.4 [-1.2 to 8.1]
  9.0: number analyzed (Participants) | 55 | 56
  9.0 | -0.8 [-5.8 to 4.2] | -1.3 [-6.5 to 4]
  12.0: number analyzed (Participants) | 61 | 60
  12.0 | 2.7 [-2.3 to 7.7] | 0.4 [-5.2 to 6.1]

50. Other Pre Specified Outcome: SF-36 Social Functioning Score
Description: SF-36 is a standardized survey evaluating 8 domains of functional health and wellbeing: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for social functioning domain was an average of the individual question scores of this domain, which are scaled 0-100 (100=highest level of functioning). The outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 0.5 Months (2 Weeks) and 3, 6, 9, and 12 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
units on a scale
  0.5: number analyzed (Participants) | 69 | 63
  0.5 | 10.9 [5 to 16.7] | 9.1 [3.2 to 15]
  3.0: number analyzed (Participants) | 68 | 64
  3.0 | 11 [4.9 to 17.2] | 5.7 [-1.4 to 12.7]
  6.0: number analyzed (Participants) | 63 | 64
  6.0 | 11.5 [5.6 to 17.4] | 6.6 [0.1 to 13.2]
  9.0: number analyzed (Participants) | 55 | 56
  9.0 | 4.5 [-1.3 to 10.4] | 12.3 [5 to 19.5]
  12.0: number analyzed (Participants) | 61 | 60
  12.0 | 6.4 [-0.4 to 13.1] | 7.1 [0.3 to 13.8]

51. Other Pre Specified Outcome: SF-36 Emotional Role Limitations Score
Description: SF-36 is a standardized survey evaluating 8 domains of functional health and wellbeing: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for emotional role limitation domain was an average of the individual question scores of this domain, which are scaled 0-100 (100=highest level of functioning). The outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 0.5 Months (2 Weeks) and 3, 6, 9, and 12 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
units on a scale
  0.5: number analyzed (Participants) | 69 | 63
  0.5 | 16.4 [5.8 to 27] | 12.2 [0.9 to 23.5]
  3.0: number analyzed (Participants) | 68 | 64
  3.0 | 19.9 [9.1 to 30.6] | 14.6 [3 to 26.2]
  6.0: number analyzed (Participants) | 63 | 64
  6.0 | 12.7 [4.7 to 20.7] | 12.5 [0.9 to 24.1]
  9.0: number analyzed (Participants) | 55 | 56
  9.0 | 13 [1.9 to 24.2] | 7.4 [-3.3 to 18.2]
  12.0: number analyzed (Participants) | 61 | 60
  12.0 | 9.8 [1.8 to 17.8] | 13.3 [2 to 24.7]

52. Other Pre Specified Outcome: SF-36 Mental Health Score
Description: as for outcome 50
Time Frame: 0.5 Months (2 Weeks) and 3, 6, 9, and 12 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
units on a scale
  0.5: number analyzed (Participants) | 69 | 63
  0.5 | 0.2 [-3.7 to 4.1] | 5 [1.3 to 8.7]
  3.0: number analyzed (Participants) | 68 | 64
  3.0 | 0.8 [-3.1 to 4.7] | 1.8 [-3.4 to 7]
  6.0: number analyzed (Participants) | 63 | 64
  6.0 | -2 [-6.4 to 2.5] | 1 [-3.5 to 5.6]
  9.0: number analyzed (Participants) | 55 | 56
  9.0 | -2.4 [-6.5 to 1.8] | 0.6 [-4.2 to 5.5]
  12.0: number analyzed (Participants) | 61 | 60
  12.0 | -0.7 [-4.8 to 3.3] | 1.3 [-3.7 to 6.2]

53. Other Pre Specified Outcome: SF-36 Physical Composite Score
Description: SF-36 is a standardized survey evaluating 8 domains of functional health and well-being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The physical composite score is a normalized t-score which combines the all 8 domains with a mean of 50 and standard deviation of 10 (higher scores indicate greater physical function). A t-score below 50 is a good all-around cutoff for detecting physical condition (per the Ware manual). The outcome is calculated as the difference in score at 2 weeks and 3, 6, or 12 months and the score at baseline.
Time Frame: 0.5 Months (2 Weeks) and 3, 6, 9, and 12 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
T-score
  0.5: number analyzed (Participants) | 69 | 63
  0.5 | 3.9 [1.7 to 6.2] | 1.5 [-0.6 to 3.6]
  3.0: number analyzed (Participants) | 68 | 64
  3.0 | 3.1 [0.8 to 5.3] | 2.6 [0.2 to 5]
  6.0: number analyzed (Participants) | 63 | 64
  6.0 | 3 [0.7 to 5.3] | 3.1 [0.7 to 5.4]
  9.0: number analyzed (Participants) | 55 | 55
  9.0 | 1.1 [-1.6 to 3.8] | 2.2 [-0.5 to 4.9]
  12.0: number analyzed (Participants) | 61 | 60
  12.0 | 2 [-0.2 to 4.2] | 2.8 [0.5 to 5.2]

54. Other Pre Specified Outcome: SF-36 Mental Composite Score
Description: SF-36 is a standardized survey evaluating 8 domains of functional health and well-being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The mental composite score is a normalized t-score which combines the all 8 domains with a mean of 50 and standard deviation of 10 (higher scores indicate greater mental health). A t-score below 52 is a well-documented cutoff for detecting depression (per the Ware manual). The outcome is calculated as the difference in score at 3, 6, or 12 months and the score at baseline.
Time Frame: 0.5 Months (2 Weeks) and 3, 6, 9, and 12 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
T-score
  0.5: number analyzed (Participants) | 69 | 63
  0.5 | 2.2 [0 to 4.5] | 3.5 [1.2 to 5.8]
  3.0: number analyzed (Participants) | 68 | 64
  3.0 | 2.7 [0.1 to 5.4] | 1.9 [-0.8 to 4.5]
  6.0: number analyzed (Participants) | 63 | 64
  6.0 | 1.6 [-0.8 to 3.9] | 1.2 [-1.2 to 3.6]
  9.0: number analyzed (Participants) | 55 | 55
  9.0 | 0.6 [-1.9 to 3.1] | 1 [-1.8 to 3.7]
  12.0: number analyzed (Participants) | 61 | 60
  12.0 | 0.9 [-1.3 to 3.1] | 1.2 [-1.7 to 4.1]

55. Other Pre Specified Outcome: Postvoid Residual Volume
Description: Postvoid Residual Volume
Time Frame: Baseline, 3, 6, and 12 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mL
Arm/Group | Botox A | Mid-Urethral Sling
Number analyzed (Participants) | 71 | 66
mL
  Baseline | 20.4 [14.6 to 26.3] | 22.7 [15.9 to 29.5]
  0.5: number analyzed (Participants) | 68 | 63
  0.5 | 49.4 [33.8 to 65.1] | 26.5 [19.5 to 33.5]
  3.0: number analyzed (Participants) | 67 | 61
  3.0 | 39.4 [25.0 to 53.7] | 27.2 [19.2 to 35.3]
  6.0: number analyzed (Participants) | 61 | 60
  6.0 | 31.7 [19.2 to 44.2] | 37.1 [23.9 to 50.3]

ADVERSE EVENTS:
Time Frame: 12 Months
Arm/Group | Botox A | Mid-Urethral Sling
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/69
Serious Adverse Events (participants affected / at risk) | 3/71 | 8/69
Other Adverse Events (participants affected / at risk) | 40/71 | 41/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Botox A (N=71) | Mid-Urethral Sling (N=69)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Botox A (N=71) | Mid-Urethral Sling (N=69)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Defaecation urgency (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyschezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Levator syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Medical device site erosion (General disorders) | 0 (0) | 2 (2)
Oedema (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Suprapubic pain (General disorders) | 0 (0) | 2 (2)
Multiple allergies (Immune system disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Coronavirus infection (Infections and infestations) | 4 (4) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 2 (2)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gonococcal pelvic inflammatory disease (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa fungal (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1)
Skin candida (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 24 (31) | 26 (34)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Biopsy breast (Investigations) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1)
Residual urine volume (Investigations) | 3 (3) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 3 (3) | 6 (6)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspareunia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic discomfort (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia areata (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Contraindication to vaccination (Social circumstances) | 0 (0) | 1 (1)
Cataract operation (Surgical and medical procedures) | 0 (0) | 1 (2)
Eye operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Spinal nerve stimulator removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1)
Vaginal mesh removal surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/31/NCT04171531/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-08): https://cdn.clinicaltrials.gov/large-docs/31/NCT04171531/SAP_001.pdf
  • Informed Consent Form (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/31/NCT04171531/ICF_002.pdf